CLINICAL TRIAL: NCT02695394
Title: Emotional Processing in Multiple Sclerosis / Clinically Isolated Syndrome: A Neuropsychological fMRI-study
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, PD Dr. Thomas Hälbig, MD, Charite University, Berlin, Germany
Other Study IDs: EA1/126/15
Record Dates: First submitted 2016-02-11; First posted 2016-03-01 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis (MS); Clinically Isolated Syndrome (CIS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MS / CIS
- Healthy controls

SUMMARY:
The aim of this prospective non-interventional neuropsychological one visit study involving functional MRI (fMRI) is to ascertain emotional processing in patients with Multiple Sclerosis (MS) or Clinically Isolated Syndrome (CIS) compared to healthy control subjects.

In different experiments, the modulation of cognitive and motor responses by visual emotional information and the ability to discriminate visual emotional stimuli will be tested using experimental behavioral paradigms. Furthermore, functional connectivity and - using fMRI - activations of brain regions known to be involved with emotional processing will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 85 years
* Right handed
* For patients: Diagnosis of CIS or diagnosis of MS since ≤5 years

Exclusion Criteria:

* Cognitive deficits as determined by a MMSE Score < 25/30
* Depression as determined by a HADS-D Score > 7
* Anxiety as determined by a HADS-A Score > 7
* Physical disabilities interfering with the study procedures or impacting outcome measures
* Clinically significant diseases within 7 days prior to the study evaluations
* Contraindications against cranial MRI without contrast

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from a academic medical center MS outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Emotional modulation of motor response time | 1 day
  Δ ([Response time following neutral stimuli] - [Response time following emotional stimuli])
Emotional memory performance | 1 day
  %-correct recognized emotional and neutral stimuli
Emotional experience | 1 day
  Subjective valence and arousal ratings of emotional and neutral stimuli

SECONDARY OUTCOMES:
BOLD-fMRI brain responses during emotional processing | 1 day
Expanded Disability Status Scale (EDSS) | 1 day
Multiple Sclerosis Functional Composite (MSFC) | 1 day
Short Form Health Survey (SF-36) | 1 day
Satisfaction With Life Scale (SWLS) | 1 day
Paced Auditory Serial Addition Test (PASAT) | 1 day
Serial Reaction Time (SRT) Task | 1 day
Symbol Digit Modalities Test (SDMT) | 1 day
Beck depression inventory BDI-2 | 1 day
Positive and Negative Affect Schedule (PANAS) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, MD, Principal Investigator — Charité Unversitätsmedizin Berlin, NeuroCure Clinical Research Center NCRC; Thomas D. Hälbig, MD, Principal Investigator — Charité Unversitätsmedizin Berlin, NeuroCure Clinical Research Center NCRC
Locations (1):
- Charité Unversitätsmedizin Berlin; NeuroCure Clinical Research Center NCRC, Berlin, Germany

REFERENCES:
- [Result] Halbig TD, Wustenberg T, Giess RM, Kunte H, Bellmann-Strobl J, Ruprecht K, Paul F. Emotional experience in patients with clinically isolated syndrome and early multiple sclerosis. Eur J Neurol. 2020 Aug;27(8):1537-1545. doi: 10.1111/ene.14269. Epub 2020 Jun 12. PMID 32307769